CLINICAL TRIAL: NCT05809765
Title: Effect of Triflow Breathing Training on Heart Rate Variability, Anxiety and Quality of Life in Hemodialysis Patients : A Randomized Control Trial
Brief Title: Effect of Triflow Breathing Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Principal Investigator, Chii Jeng, Professor, Taipei Medical University WanFang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: N202001049
Record Dates: First submitted 2023-03-09; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Hemodialysis Complication; Haemolyses and Related Conditions
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Intervention Model Description: The participants were divided into the first group of patients undergoing hemodialysis every Monday, Wednesday, and Friday and the second group undergoing dialysis every Tuesday, Thursday, and Saturday. The experimental group and the control group were randomly assigned by a coin toss. The investigators conducted the study for eight weeks and investigated the effects of respiration training on the improvement of heart rate variability, anxiety, and quality of life in hemodialysis patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 dialysis on Mondays, Wednesdays, and Fridays (Other): 8-week breath training by using a disposable, flow-oriented, Triflow three-ball incentive spirometer.
  Interventions: Other: 8-week breath training program
- Group 2 dialysis on Tuesdays, Thursdays, and Saturdays (Other): 8-week breath training by using a disposable, flow-oriented, Triflow three-ball incentive spirometer.
  Interventions: Other: 8-week breath training program

INTERVENTIONS:
Other: 8-week breath training program — The participants were asked to be seated comfortably and raise their heads by 30° with the guidance of the investigator. During the inspiration process, the participants' abdomens bulged. They then held their breaths for 5 seconds before exhaling from their mouths for twice the duration of inspiration. Breath training was performed five times each hour throughout the three-hour duration of each dialysis session. In sum, the experimental group performed Triflow breath training 15 times during each dialysis session. The experimental group and the control group were randomly assigned by a coin toss.

SUMMARY:
This study aims to explore whether an 8-week Triflow breath training program reduced the anxiety levels and improved the heart rate variability and quality of life of patients receiving hemodialysis. To investigate the effect of the triflow respiration training on the improvement of heart rate variability, anxiety, and the quality of life in hemodialysis patients.

DETAILED DESCRIPTION:
Method:This research adapted the cluster randomization design. The participants were divided into the first group of patients undergoing hemodialysis every Monday, Wednesday, and Friday and the second group undergoing dialysis every Tuesday, Thursday, and Saturday. The experimental group and the control group were randomly assigned by a coin toss. The investigators conducted the study for eight weeks and investigated the effects of respiration training on the improvement of heart rate variability, anxiety, and quality of life in hemodialysis patients. Patients in the experimental group receive the triaflow respiration training three times a week for eight weeks during hemodialysis. Data were collected by a heart rate variability monitor, State-Trait Anxiety Inventory and WHOQOL-BREF at baseline and after a 8-week respiration training.

ELIGIBILITY:
Inclusion Criteria:

1. Long-term hemodialysis is required to treat patients with end-stage renal disease diagnosed by a physician.
2. Blood older than or equal to 65 years old and under 80 years old with diabetes Dialysis patients.
3. Hemodialysis has been accepted for more than three months and is still under treatment and half There were no hospitalizations for other comorbidities during the year.
4. Those who are conscious and have no serious mental symptoms, can talk and express and agree to Subject to respirator training and questionnaires.
5. Available country and Taiwanese communicators.
6. The average score of the Situational Trait Anxiety Scale is greater than 20 points.

Exclusion Criteria:

1. Patients with low blood pressure during dialysis can not raise the bed to 30 degrees.
2. Blindness and hearing or long-term bedridden.
3. There are cases of irregular heartbeat.
4. The Daily Activity Scale is less than or equal to 60 points (the study uses the Barthel Index).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-05-16 (Actual); Primary Completion 2021-05-14 (Actual); Study Completion 2021-05-14 (Actual)

PRIMARY OUTCOMES:
Changes of heart rate variability, the measurement indices were the total power, which reflects the autonomic tone; the low-frequency component of heart rate variability. | For the experimental group, heart rate variability was measured each week during the 8-week breath training. For the control group, heart rate variability was measured at the first, 4th and the 8th week.
  The heart rate variability was measured using the 60601-1 program provided by Daily Care BioMedical, and the balance of their autonomic nervous systems was analyzed using the 60601-1 software.
Changes of the level of anxiety | The level of anxiety was measured at the first week, 4th week and the 8th week.
  The State-Trait Anxiety Inventory (STAI) is used to measure the levels of anxiety. It consists of two subscales: one for state anxiety and the other for trait anxiety. Each subscale comprises 20 items, rated using a 4-point Likert scale (1 = hardly; 2 = sometimes; 3 = often; and 4 = almost always), with a total score of 20-80.
Changes of the level of quality of life | The level of quality of life was measured at the first week, 4th week and the 8th week.
  The Chinese version of World Health Organization Quality of Life Brief Edition (WHOQoL-BREF) was used, which consists of 28 items. All items are rated using a 5-point Likert scale. Each Quality of life dimension differs in the number of items, and its score is determined by multiplying the mean score of all its items by 4. The average score of each dimension ranges from 4 to 20, with a higher score indicating a better Quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Chii Jeng, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No